CLINICAL TRIAL: NCT02425384
Title: Accelerometer-linked Online Intervention to Promote Physical Activity in Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HopeLab Foundation (Other)
Collaborators: West Virginia University (Other); Santech, Inc (Industry); Stanford University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: HL-GD001
Record Dates: First submitted 2015-04-16; First posted 2015-04-24 (Estimated); Last update posted 2015-04-24 (Estimated); Status verified 2015-04

CONDITIONS: Health Behavior; Adolescent Behavior; Motivation
Keywords: adolescent; physical activity; accelerometer
MeSH Terms: conditions — Health Behavior; Adolescent Behavior; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Intervention Group (Experimental): This group is provided an activity meter that tracks the amount and intensity of one's physical activity and is linked to a motivational website. On the website, activity data from the activity meter can be viewed after uploading information from the meter to the website. The reward website allots points for participants based on the amount and intensity of physical activity. Points can be redeemed for rewards on the website, such as gift cards and digital badges.
  Interventions: Behavioral: Intervention Group (motivational website, activity meter)
- Active Control (Active Comparator): This group is provided an activity meter that tracks the amount and intensity of one's physical activity and a copy of the game Dance Dance Revolution (DDR). The activity meter will upload data to a secure server but will not be linked to the motivational website used by the intervention group. DDR is a dancing video game in which players view arrows timed to music on a TV screen and gain points by stepping on the corresponding arrows on a floor mat. Players obtain points in the game by stepping on the correct arrows at the right time to the beat of the music. The points earned with DDR cannot be redeemed for rewards.
  Interventions: Behavioral: Active Control (active video game, activity meter)
- Passive Control (Placebo Comparator): This group is provided with an activity meter and will be asked to carry it with them as they go about their normal daily activities. Like in the Active Control group, participants in the Passive Control group will not have access to the motivational website. For this group, the activity meter functions solely as a monitor to track their activity levels. No other product or intervention will be introduced to the control group.
  Interventions: Other: Passive Control (activity meter)

INTERVENTIONS:
Behavioral: Intervention Group (motivational website, activity meter) — The activity meter linked to a motivational website is designed to motivate middle school-aged children to increase their rates of physical activity by providing feedback on the amount of activity, and rewards based on the amount and duration of activity.
  Arms: Intervention Group
Behavioral: Active Control (active video game, activity meter) — The active video game, Dance Dance Revolution, requires physical movement as part of game play and may motivate users to engage in more activity. The same activity meter used in the Intervention Group is provided to this group to track physical activity but does not link to the motivational website nor does it provide any feedback on levels or duration of activity.
  Arms: Active Control
Other: Passive Control (activity meter) — Participants are provided the same activity meter used in the other study groups to track physical activity but it does not link to the motivational website nor does it provide any feedback on levels or duration of activity. Participants are asked to go about their normal activities.
  Arms: Passive Control

SUMMARY:
The primary objective of this protocol is to test whether an activity monitor with an online motivational rewards component will increase physical activity levels of middle school-aged students. The secondary objective is to learn about the functionality and utilization of the activity meter device among this age group.

DETAILED DESCRIPTION:
The goal of this pilot study is to find out whether an activity meter linked to web-based rewards will increase physical activity levels in middle school aged students who use it over 6 weeks. To test this, students who participate in the study will be assigned to 1 of 3 groups: the meter with web-based rewards group, the Dance Dance Revolution group, or the control group. The physical activity of participants in all 3 groups will be tracked using the an activity meter that participants will be asked to carry daily for the 6 weeks of the study. Participants given the activity meter with web-based rewards or Dance Dance Revolution will be instructed to use them at their own will, as much or as little as they like. Before beginning the study, all participating students will be asked background questions about themselves (such as their gender, age, and ethnic group) and about the kinds of computer and video game consoles they have access to at home. All participants will also complete short questionnaires at enrollment, week 1, week 3 and week 6. These questions will ask participants about their experiences using the assigned devices, their physical activity levels, and their thoughts about their ability to be physically active. At the end of 6 weeks, all participants will finish the study and return their assigned devices to the study coordinator. Height and weight will be measured at baseline and at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Any student 11 to 14 years old with access to a computer that uses either Windows XP or Mac OS X 10.4 operating system with internet access.

Exclusion Criteria:

* Anyone with a medical condition or existing health complications that will interfere with their ability to be physically active.
* Inability to read and write English (though consent forms for parents that speak other languages will be provided).

Ages: 11 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 182 (Actual)
Dates: Start 2008-10; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Physical Activity | 6 weeks
  The amount and intensity of physical activity is recorded continuously every study day that participants wear the provided activity meter for the 6 weeks study. The primary outcome reported will be rates of "moderate to vigorous" physical activity.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Cole, PhD, Principal Investigator — HopeLab Foundation
Locations (3):
- United States (3):
  - Crittenden Middle School, Mountain View, California
  - Vista Middle School, Vista, California
  - West Virginia University, Morgantown, West Virginia